CLINICAL TRIAL: NCT04325113
Title: Post Tonsillectomy Analgesia Comparison After Surgery Site Spray of NaCl 0,9%, Xylocaine 2% or Levobupivacaine 0,5%
Brief Title: Post Tonsillectomy Analgesia Comparison After Surgery Site Spray of Local Anesthesics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tonsilstopic
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Levobupivacaine; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NaCl 0,9% (Placebo Comparator): patients receive 5ml of NaCl 0,9% at the level of the tonsils lodge
  Interventions: Drug: levobupivacaine
- Xylocaine 2% (Active Comparator): patients receive 5ml of Xylocaïne 2% at the level of the tonsils lodge
  Interventions: Drug: levobupivacaine
- Levobupivacaine 0,5% (Active Comparator): patients receive 5ml of Levobupivacaine 0,5% at the level of the tonsils lodge
  Interventions: Drug: levobupivacaine

INTERVENTIONS:
Drug: levobupivacaine — Patient satisfaction and pain score using a visual anagogic scale (VAS)
  Other Names: xylocaine; Nacl

SUMMARY:
Check analgesia after tonsillectomy in adults

DETAILED DESCRIPTION:
We hypothesize that a vaporization of local anesthetics in the tonsil lodge would reduce postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Tonsillectomy

Exclusion Criteria:

* Gastric or duodenal ulcer
* Diabetes
* Kidney failure
* Chronic pain and fibromyalgia

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction and pain score | until 10 days after the tonsillectomy.
  patient satisfaction and pain score using a visual anagogic scale from 0 (no pain) to 10 (intolerable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Javillier, Liège, Belgium